CLINICAL TRIAL: NCT06857487
Title: Efficacy and Safety of Qingre Huatan Formula for the Prevention of Early Neurological Deterioration in Patients With Acute Ischemic Stroke : A Randomized Double-blind Placebo-controlled Pilot Trial
Brief Title: Qingre Huatan Formula for the Prevention of Early Neurological Deterioration in Acute Ischemic Stroke
Acronym: QUIET
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023DZMEC-410-02
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qingre Huatan Formula (Experimental): Patients will receive orally administered Qingre Huatan Formula, combined with guidelines-based standard care.
  Interventions: Drug: Qingre Huatan Formula; Other: Guidelines-based standard care
- Qingre Huatan Formula placebo (Placebo Comparator): Patients will receive orally administered Qingre Huatan Formula placebo, combined with guidelines-based standard care.
  Interventions: Drug: Qingre Huatan Formula placebo; Other: Guidelines-based standard care

INTERVENTIONS:
Drug: Qingre Huatan Formula — Qingre Huatan Formula, granules, 1 bag each time, twice a day, orally, continue for 10 days.
  Arms: Qingre Huatan Formula
Drug: Qingre Huatan Formula placebo — Qingre Huatan Formula placebo, granules, 1 bag each time, twice a day, orally, continue for 10 days.
  Arms: Qingre Huatan Formula placebo
Other: Guidelines-based standard care — Guidelines-based standard care for acute ischemic stroke

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of Qingre Huatan formula versus placebo on preventing early neurological deterioration in patients with acute ischemic stroke within 48 hours after onset.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients diagnosed with acute ischemic stroke. Inpatients diagnosed of acute ischemic stroke.
2. Meet the criteria of TCM phlegm-heat syndrome
3. Patients at high-risk of END : Magnetic resonance imaging (MRI) reveals new ischemic lesions, with DWI-ASPECTS score ≤ 7, or presence of at least two risk factors of END.
4. Acute ischemic stroke within 48 hours after onset.
5. Aged 18-80 years, male or female.
6. The patient or representative has signed informed consent.

Exclusion Criteria:

1. Received or planned thrombolysis or endovascular therapy after onset.
2. Suspected secondary stroke caused by brain tumor, brain trauma, hemopathy, etc.
3. Already dependent in activities of daily living before the present acute stroke (defined as modified Rankin Scare score ≥2 )
4. Diseases that cause motor dysfunction, including osteoarthritis, etc.
5. Known severe liver or kidney dysfunction (alanine aminotransferase or aspartate transaminase > 2 times the upper limit of normal value, serum creatinine > 1.5 times the upper limit of normal value)
6. Known severe aphasia or mental illness affecting clinical information collection and evaluation.
7. Pregnancy, potential pregnancy or breastfeeding.
8. Currently participating in other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-10-24 (Estimated); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
The incidence of early neurological deterioration within 7 days of onset | Basline and Day 7
  An increase of NIHSS ≥2 within 7 days of onset is considered as early neurological deterioration. The NIHSS (National Institute of Health Stroke Scale) is a neurological assessment tool for stroke patients, with scores ranging from 0 to 42.

SECONDARY OUTCOMES:
Change in National Institute of Health Stroke Scale scores from baseline to 10 days (after the treatment) | Basline and 10 days after treatment initiation
  The NIHSS (National Institute of Health Stroke Scale) is a neurological assessment tool for stroke patients, with scores ranging from 0 to 42. Scores of 0-1 indicate near normal status, 1-4 mild stroke, 5-15 moderate stroke, 16-20 moderate-to-severe stroke, and 21-42 severe stroke. It is primarily used to quickly assess stroke severity and guide treatment decisions.
The proportion of patients with modified Rankin Scale score ≤2 on day 30 | Day 30
  The mRS (modified Rankin Scale) is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranging from 0 (no symptom) to 5 (severe disability) and 6 (death).
The proportion of patients with modified Rankin Scale score ≤2 on day 90 | Day 90
  The mRS (modified Rankin Scale) is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranging from 0 (no symptom) to 5 (severe disability) and 6 (death).
Activity of daily living of patients measured by Barthel Index score on day 30 | Day 30
  Barthel Index is a commonly used scale for measuring the activity of daily living of people. Score of 10-item scale ranges from 0 (worst) to 100 (best).
Activity of daily living of patients measured by Barthel Index score on day 90 | Day 90
  Barthel Index is a commonly used scale for measuring the activity of daily living of people. Score of 10-item scale ranges from 0 (worst) to 100 (best).
Incidence of treatment-related adverse events | 90 days after treatment initiation
  Number of patients with any adverse events during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China